CLINICAL TRIAL: NCT03989570
Title: Ultrasound Guided Transversus Abdominis Plane Block Versus Erector Spinae Plane Block in Patients Undergoing Emergency Laparotomies.
Brief Title: Transversus Abdominis Plane Block Versus Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hassan Mokhtar Elshorbagy Hetta (Other)
Responsible Party: Sponsor-Investigator, Hassan Mokhtar Elshorbagy Hetta, assistant lecture, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 73-7/2018
Record Dates: First submitted 2019-05-04; First posted 2019-06-18 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain; Laparotomy
Keywords: Erector Spinae Plane Block; Transversus Abdominis Plane Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (A group) (Experimental): 31 patients Will undergo ESP block with 40 ml bupivacine 0.25% (20 ml on each side), and TAP block with 40 ml saline 0.9% (20 ml on each side).
  Interventions: Procedure: erector spinae plane block
- Group II (B group) (Active Comparator): 31patients Will undergo TAP block with 40 ml bupivacine 0.25% (20 ml on each side), and ESP block with 40 ml saline 0.9% (20 ml on each side).
  Interventions: Procedure: transversus abdominis plane block
- Group III (C group) (Placebo Comparator): 31 patients anesthetized with the protocol followed by Minia University Hospital
  Interventions: Other: control group

INTERVENTIONS:
Procedure: transversus abdominis plane block — The TAP block will be performed laterally behind the midaxillary line between the iliac crest and the most inferior extent of the ribs. The plane between the internal oblique and transversus abdominis muscle will be located around the midaxillary line with the probe transverse to the abdomen. Anteriorly,The needle will be passed to come in plane with the ultrasound beam and placed between transversus and internal oblique posterior to the midaxillary line then, the local anesthetic will be injected
  Arms: Group II (B group)
Procedure: erector spinae plane block — The ESP block will be performed into a fascial plane between the deep surface of erector spinae muscle and the transverse processes
  Arms: Group I (A group)
Other: control group — placebo
  Arms: Group III (C group)

SUMMARY:
The TAP block, first described by Rafi in 2001, is comprised of deposition of a local anesthetic into the anatomical plane between the internal oblique and transverses abdominis muscles, where thess thoracoabdominal nerves (T6-L1) contribute to the main sensory supply of the skin, muscles, and parietal peritoneum of the anterior abdominal wall. These nerves branch and communicate extensively with each other in the TAP .

Erector spinae plane (ESP) block is a recently described interfascial block in which the local anaesthectic is placed over or below the plane of the erector spinae muscle, near where the spinal nerves come out from the spine before they start to divide. Some publications have shown its effectiveness in treating thoracic and abdominal postoperative pain.

Postoperative pain is the major obstacle for early postoperative ambulation and increases the risk of venous thromboembolism, respiratory complications and prolongs the hospital stay. Parietal pain is the chief component of postoperative pain after abdominal surgeries. Large doses of opioids are required to mitigate this pain, but they are poorly tolerated. Multimodal analgesia is effective in handling postoperative pain and in attenuating the side effects of large doses of a single analgesic .

DETAILED DESCRIPTION:
Group I (A group): Will undergo ESP block with 40 ml bupivacine 0.25% (20 ml on each side), and TAP block with 40 ml saline 0.9% (20 ml on each side).

Group II (B group): Will undergo TAP block with 40 ml bupivacine 0.25% (20 ml on each side), and ESP block with 40 ml saline 0.9% (20 ml on each side).

Group III (C group): anesthetized with the protocol followed by Minia University Hospital The medication will be prepared and supplied in similar syringes by an anesthetist not included in the management of the patint or data collection.

Methods:

Following placement of the standard monitors, intravenous access will secured and the patients will started on IV fluids. Anesthesia will be induced with 0.04 mg/kg midazolam, 2 μg/kg fentanyl, and titrated doses of propofol. Endotracheal intubation will facilitated with 0.5 mg/kg of atracurium. Isoflurane 1.2%, will be used for anesthetic maintenance After induction of anesthesia, stabilizing the patient's hemodynamics, and before surgical incision, ESB & TAP block will be performed. With the patient in the supine position, the site of the ultrasound and needle entry will be sterilized. The TAP block will be performed laterally behind the midaxillary line between the iliac crest and the most inferior extent of the ribs. The plane between the internal oblique and transversus abdominis muscle will be located around the midaxillary line with the probe transverse to the abdomen. Anteriorly,The needle will be passed to come in plane with the ultrasound beam and placed between transversus and internal oblique posterior to the midaxillary line then, the local anesthetic will be injected. Then the patient will turn in lateral position, the site of the ultrasound and needle entry will be sterilized. The ESP block will be performed into a fascial plane between the deep surface of erector spinae muscle and the transverse processes

ELIGIBILITY:
Inclusion Criteria:

* 1. Age18-70 . 2. Both gender . 3 .Emergency laparotomies . 4. ASA I-III .

Exclusion Criteria:

1. Drug allergy .
2. Morbid obesity (BMI >40 kg/m2) .
3. Psychiatric disorder .
4. Opioid dependence .
5. patient refuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagy S. Ali, MD, Study Chair — Minia University Hospital; Abeer A Hassanien, Study Director — Minia University Hospital
Locations (1):
- Minia University Hospital, Minya, Egypt

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 patient refuse to participate
Period: Overall Study
Arm/Group | Group I (A Group) | Group II (B Group) | Group III (C Group)
Started | 31 | 31 | 31
Completed | 31 | 31 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (A Group) | Group II (B Group) | Group III (C Group) | Total
Number analyzed (Participants) | 31 | 31 | 31 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (14.9) | 47.4 (11.8) | 43.6 (13.7) | 45.61 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 16 | 45
  Male | 16 | 17 | 15 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 31 | 31 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 31 | 31 | 31 | 93
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 31 | 31 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Time of First Post Operative Analgesic Request
Description: the pain will be assisted based on the time for the first dose of rescue analgesia
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Group I (A Group) | Group II (B Group) | Group III (C Group)
Number analyzed (Participants) | 31 | 31 | 31
Hour | 14.9 (5.7) | 6.5 (2.2) | 2.8 (1.6)

2. Primary Outcome: Postoperative Total Fentanyl Requirement
Description: The total amount of postoperative fentanyl in milligram was given to the patient as rescue analgesia during 24 hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | Group I (A Group) | Group II (B Group) | Group III (C Group)
Number analyzed (Participants) | 31 | 31 | 31
Milligram | 40.3 (26.7) | 111 (38.1) | 175 (38.9)

3. Secondary Outcome: Incidence of Any Adverse Events
Description: adverse events related to technique or drugs
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Group I (A Group) | Group II (B Group) | Group III (C Group)
Number analyzed (Participants) | 31 | 31 | 31
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 days
Description: All patients were under control and receive the best care of management Our techniques don't make any side effects or affect patients outcome
Arm/Group | Group I (A Group) | Group II (B Group) | Group III (C Group)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT03989570/Prot_SAP_000.pdf